CLINICAL TRIAL: NCT02152293
Title: Pharmacoepidemiology Study on Real Life Impact of Chloroprocaine (CLOROTEKAL®) on the Eligibility for Discharge From Hospital of Patients Requiring Short Outpatient Surgery Under Spinal Anesthesia
Brief Title: Impact of Chloroprocaine (CLOROTEKAL®) on Eligibility for Discharge From Hospital After Outpatient Surgery
Acronym: CLOCK
Status: Completed | Type: Observational
Sponsor: Nordic Pharma SAS (Industry)
Responsible Party: Sponsor
Other Study IDs: CLOCK
Record Dates: First submitted 2014-05-23; First posted 2014-06-02 (Estimated); Last update posted 2015-05-25 (Estimated); Status verified 2015-05

CONDITIONS: Spinal Anesthesia; Outpatient Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to assess, in real life, the efficacy and the eligibility for discharge of a local anesthetic, CLOROTEKAL®, used for spinal anesthesia in short outpatient surgery.

DETAILED DESCRIPTION:
This is a longitudinal, observational, prospective, multicentre, national study, conducted in France, from a representative sample of physician anesthetists.

The efficacy and safety in real life of CLOROTEKAL® will be assessed in patients undergoing a short outpatient surgery under spinal anesthesia. Data will be collected by the physician during two visits (pre-anesthesia and per-postoperative consultation). Additional data regarding the patient's perception (safety, pain and satisfaction) will be collected using a self-questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients seen in pre-anesthesia consultation for ambulatory surgery
* Patients for whom a spinal anesthesia using CLOROTEKAL® is planned
* Patients accepting and able to complete a satisfaction self-administered questionnaire
* Informed patients who accept the computer processing of their medical data and their right of access and correction

Exclusion Criteria:

* Patients with contra-indications to spinal anesthesia (eg decompensated cardiac insufficiency, hypovolemic shock….)
* Patients with contra-indications to chloroprocaine (hypersensitivity to the active substance, medicinal products of the para-aminobenzoic acid ester group, other ester-type local anaesthetics or to any of the excipients ; Intravenous regional anaesthesia (the anesthetic agent is introduced into the limb and allowed to set in while tourniquets retain the agent within the desired area), serious problems with cardiac conduction, severe anemia)
* Patients participating or having participated in the previous month in a clinical trial in anesthesiology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for surgery under spinal anesthesia of short duration will be informed about the study and will be asked to participate, from about day -14 (pre-anesthesia consultation) to 24h after the day of surgery.
Sampling Method: Non-Probability Sample
Enrollment: 620 (Actual)
Dates: Start 2014-05; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Impact of CLOROTEKAL® on the discharge from hospital | Average time expected around 180 min after the surgery (Lacasse, 2011)
  Time to eligibility for discharge from hospital measured as the time between the intrathecal injection and achieving the criteria of Lacasse.
  This period will be described globally (average time) and by groups: <180 min ; <240 min ; <300 min ; <360 min ; > 360 min.

SECONDARY OUTCOMES:
Modalities of spinal anesthesia with CLOROTEKAL® | During surgery
Safety of CLOROTEKAL | Up to 24 hours after surgery
  Percentage and nature of adverse effect (serious or not) after intrathecal anaesthesia with chloroprocaine.
Patients' satisfaction | 24h after surgery
Postoperative patients pain | During the 24 hours following surgery
Rate of unplanned admissions related to anesthesia and/or surgery | Within the same day than surgery

CONTACTS AND LOCATIONS:
Overall Officials: Hélène HERMAN-DEMARS, MD, Study Director — Nordic Pharma
Locations (1):
- Nordic Pharma, Paris, France

REFERENCES:
- [Background] Lacasse MA, Roy JD, Forget J, Vandenbroucke F, Seal RF, Beaulieu D, McCormack M, Massicotte L. Comparison of bupivacaine and 2-chloroprocaine for spinal anesthesia for outpatient surgery: a double-blind randomized trial. Can J Anaesth. 2011 Apr;58(4):384-91. doi: 10.1007/s12630-010-9450-x. Epub 2011 Jan 4. PMID 21203878
- [Derived] Capdevila X, Aveline C, Delaunay L, Bouaziz H, Zetlaoui P, Choquet O, Jouffroy L, Herman-Demars H, Bonnet F. Impact of Chloroprocaine on the Eligibility for Hospital Discharge in Patients Requiring Ambulatory Surgery Under Spinal Anesthesia: An Observational Multicenter Prospective Study. Adv Ther. 2020 Jan;37(1):541-551. doi: 10.1007/s12325-019-01172-5. Epub 2019 Dec 11. PMID 31828611